CLINICAL TRIAL: NCT03692910
Title: A 2-Part Study (Open-label Followed by Double-blind, Randomized, Placebo-controlled, Parallel Group) of the Safety, Tolerability, Pharmacokinetics, and Efficacy of SAGE-217 in the Treatment of Subjects With Bipolar I/II Disorder With a Current Major Depressive Episode
Brief Title: A Study to Evaluate SAGE-217 in Participants With Bipolar I/II Disorder With a Current Major Depressive Episode
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 217-BPD-201
Record Dates: First submitted 2018-09-12; First posted 2018-10-02 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Bipolar Disorder I; Bipolar Disorder II; Major Depressive Episode
MeSH Terms: conditions — Bipolar Disorder | interventions — zuranolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Open-label): SAGE-217 (Experimental): Participants self-administered SAGE-217, 30 milligrams (mg), oral capsule, once daily (QD), in the evening, from Day 1 to Day 14.
  Interventions: Drug: SAGE-217
- Part B (Double-blind): SAGE-217 (Experimental): Participants were to receive SAGE-217, 30 mg, oral capsule, QD, in the evening, from Day 1 to Day 14 in Part B of the study. However, as per the Sponsor's decision, the Part B of the study was not conducted.
  Interventions: Drug: SAGE-217
- Part B (Double-blind): Placebo (Placebo Comparator): Participants were to receive SAGE-217 matching placebo capsule, orally, QD, in the evening, from Day 1 to Day 14 in Part B of the study. However, as per the Sponsor's decision, the Part B of the study was not conducted.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAGE-217 — SAGE-217 capsule
  Arms: Part A (Open-label): SAGE-217; Part B (Double-blind): SAGE-217
Drug: Placebo — SAGE-217 matching placebo capsule
  Arms: Part B (Double-blind): Placebo

SUMMARY:
This is an open-label study evaluating the safety, tolerability, pharmacokinetics, and efficacy of SAGE-217 in the treatment of participants with bipolar I/II disorder with a current major depressive episode.

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

1. Participant had a documented history of hypomanic or manic episode and a diagnosis of bipolar I or bipolar II disorder with a current major depressive episode.

Exclusion Criteria:

1. Participant had a history of suicide attempt.
2. Participant had current suicidal ideation with plans.
3. Participant had a history of rapid cycling bipolar disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-05-21 (Actual); Study Completion 2019-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Sage Investigational Site, Little Rock, Arkansas
  - Sage Investigational Site, Garden Grove, California
  - Sage Investigational Site, Lemon Grove, California
  - Sage Investigational Site, Orange, California
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Lauderhill, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, St Louis, Missouri
  - Sage Investigational Site, Austin, Texas
  - Sage Investigational Site, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 11 investigative sites in the United States from 23 August 2018 to 21 May 2019.
Pre-assignment Details: The study was to be conducted in 2 parts: Part A (Open-label) and Part B (Double-blind). Participants received SAGE-217 during the treatment period in Part A. Part B was to be initiated post review of Part A data. However, as per the Sponsor's decision, Part B was not conducted and hence no participants were enrolled in it and no data collection and analysis was done.
Period: Overall Study
Arm/Group | Part A (Open-label): SAGE-217 | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Started | 35 | 0 | 0
Completed | 29 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received at least one dose of study drug.
Groups:
- Part A (Open-label): SAGE-217: Participants self-administered SAGE-217, 30 mg, oral capsule, QD, in the evening, from Day 1 to Day 14.
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With at Least One Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE was defined as an adverse event with onset after the start of study through Day 42/early termination.
Time Frame: From first dose of study drug up to Day 42
Population: Safety Set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 35
Participants | 16

2. Primary Outcome: Part A: Number of Participants With TEAEs, Graded by Severity
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE was defined as an adverse event with onset after the start of study through Day 42/early termination. Severity was assessed according to the following scale: mild (awareness of sign or symptom, but easily tolerated); moderate (discomfort sufficient to cause interference with normal activities); severe (incapacitating, with inability to perform normal activities).
Time Frame: From first dose of study drug up to Day 42
Population: Safety Set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 35
Participants
  Mild | 11
  Moderate | 5
  Severe | 0

3. Primary Outcome: Part A: Percentages of Participants With Response to Suicidal Ideation and Suicidal Behavior Based on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Suicidality was monitored using the C-SSRS. This scale consists of a baseline evaluation that assesses the lifetime experience of the participant with suicidal ideation and behavior, and a post-baseline evaluation that focuses on suicidality since the last study visit. The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) and behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt (non-fatal), completed suicide). Percentage of participants with response 'yes' are reported for both suicidal ideation and behavior.
Time Frame: Baseline, Post-baseline (any time up to Day 42)
Population: Safety Set included all participants who received at least one dose of study drug. Number analyzed is the number of participants with data available for analyses at the specific time point.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 35
percentage of participants
  Suicidal Ideation: Baseline | 22.9
  Suicidal Ideation: Post-Baseline (Any Time up to Day 42): number analyzed (Participants) | 32
  Suicidal Ideation: Post-Baseline (Any Time up to Day 42) | 9.4
  Suicidal Behavior: Baseline | 0
  Suicidal Behavior: Post-Baseline (Any Time up to Day 42): number analyzed (Participants) | 32
  Suicidal Behavior: Post-Baseline (Any Time up to Day 42) | 0

4. Primary Outcome: Part A: Change From Baseline in the Young Mania Rating Scale (YMRS) Total Score
Description: Manic symptoms were assessed during the study using the YMRS. The clinician-administered scale is based on 11 items of core symptoms of mania. Four of the items (irritability, speech, thought content, and disruptive/aggressive behavior) were graded on a scale of 0 to 8 (choices given as even numbers), with the remaining 7 items graded on a scale of 0 to 4. Scoring between the points given (whole or half points) is possible. The YMRS total score ranges from 0 (no symptoms) to 60 (extreme severity of symptoms). A higher total score indicates a greater degree of mania. A negative change indicates better state of health.
Time Frame: Baseline, Days 3, 8, 12, 15, 21, 28, 35, and 42, Last value on treatment (up to Day 14), Last value on study (up to Day 42)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 35
score on a scale
  Baseline | 4.9 (3.23)
  Change From Baseline at Day 3: number analyzed (Participants) | 30
  Change From Baseline at Day 3 | -0.9 (2.24)
  Change From Baseline at Day 8: number analyzed (Participants) | 27
  Change From Baseline at Day 8 | -0.9 (2.66)
  Change From Baseline at Day 12: number analyzed (Participants) | 26
  Change From Baseline at Day 12 | -0.7 (3.35)
  Change From Baseline at Day 15: number analyzed (Participants) | 23
  Change From Baseline at Day 15 | 0.3 (3.10)
  Change From Baseline at Day 21: number analyzed (Participants) | 29
  Change From Baseline at Day 21 | -0.7 (3.08)
  Change From Baseline at Day 28: number analyzed (Participants) | 28
  Change From Baseline at Day 28 | -0.9 (2.92)
  Change From Baseline at Day 35: number analyzed (Participants) | 29
  Change From Baseline at Day 35 | -0.9 (3.29)
  Change From Baseline at Day 42: number analyzed (Participants) | 29
  Change From Baseline at Day 42 | -1.3 (2.85)
  Change at Last Value on Treatment (up to Day 14): number analyzed (Participants) | 31
  Change at Last Value on Treatment (up to Day 14) | -0.2 (3.28)
  Change at Last Value on Study (up to Day 42): number analyzed (Participants) | 32
  Change at Last Value on Study (up to Day 42) | -1.2 (3.02)

5. Primary Outcome: Part B: Change From Baseline in the 17-Item Hamilton Depression Rating Scale (HAM-D) Total Score
Description: The 17-item HAM-D was used to rate the severity of depression in participants who were identified as experiencing a major depressive episode (MDE). Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4 include: agitation, depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), anxiety (psychic and somatic), hypochondriasis. The HAM-D total score was calculated as the sum of the 17 individual item scores, with a range of 0 (not at all depressed) to 52 (severely depressed). Higher scores indicated more depression. A negative change from baseline indicates improvement.
Time Frame: Baseline up to Day 42
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Part A: Change From Baseline in the 17-Item HAM-D Total Score at Day 15
Description: The 17-item HAM-D was used to rate the severity of depression in participants who were identified as experiencing an MDE. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4 include: agitation, depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), anxiety (psychic and somatic), hypochondriasis. The HAM-D total score was calculated as the sum of the 17 individual item scores, with a range of 0 (not at all depressed) to 52 (severely depressed). Higher scores indicated more depression. A negative change from baseline indicates improvement.
Time Frame: Baseline, Day 15
Population: Efficacy Set included all participants that received at least 1 dose of study drug, and who had at least one post-baseline Hamilton Depression Rating Scale (HAM-D) evaluation. Number analyzed is the number of participants with data available for analyses at the specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 32
score on a scale
  Baseline | 25.7 (2.97)
  Day 15: number analyzed (Participants) | 23
  Day 15 | -11.4 (8.69)

7. Secondary Outcome: Part A: Percentage of Participants With HAM-D Response at Day 15
Description: HAM-D response was defined as having a 50% or greater reduction from baseline in HAM-D total score. The HAM-D total score was calculated as the sum of the 17 individual item scores. The 17-item HAM-D comprises individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. The HAM-D total score was calculated as the sum of the 17 individual item scores, with a range of 0 (not at all depressed) to 52 (severely depressed). Higher scores indicated more depression.
Time Frame: Day 15
Population: Efficacy Set included all participants that received at least 1 dose of study drug, and who had at least one post-baseline Hamilton Depression Rating Scale (HAM-D) evaluation. Overall number of participants analyzed were the participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 23
percentage of participants | 43.5

8. Secondary Outcome: Part A: Percentage of Participants With HAM-D Remission at Day 15
Description: HAM-D remission was defined as having a HAM-D total score of ≤7. The HAM-D total score was calculated as the sum of the 17 individual item scores. The 17-item HAM-D comprises individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. The HAM-D total score was calculated as the sum of the 17 individual item scores, with a range of 0 (not at all depressed) to 52 (severely depressed). Higher scores indicated more depression.
Time Frame: Day 15
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 23
percentage of participants | 30.4

9. Secondary Outcome: Part A: Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at Day 15
Description: The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. It includes questions on the following symptoms: apparent sadness; reported sadness; inner tension; reduced sleep; reduced appetite; concentration difficulties; lassitude; inability to feel; pessimistic thoughts; and suicidal thoughts. Each item was scored in a range of 0 (no symptoms) to 6 (symptoms of maximum severity). The MADRS total score was calculated as the sum of the ten individual item scores and ranges from 0 (symptoms absent) to 60 (severe depression). Higher MADRS scores indicate more severe depression. A negative change indicates improvement.
Time Frame: Baseline, Day 15
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 32
score on a scale
  Baseline | 34.4 (4.58)
  Change From Baseline at Day 15: number analyzed (Participants) | 23
  Change From Baseline at Day 15 | -15.5 (11.67)

10. Secondary Outcome: Part A: Change From Baseline in Response to the Clinical Global Impression - Severity (CGI-S) at Day 15
Description: The CGI-S uses a 7-point Likert scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who had the same diagnosis. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=extremely ill. A negative change from baseline indicates improvement (higher absolute number indicating more illness).
Time Frame: Baseline, Day 15
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 32
score on a scale
  Baseline | 4.4 (0.62)
  Change From Baseline at Day 15: number analyzed (Participants) | 23
  Change From Baseline at Day 15 | -1.4 (1.24)

11. Secondary Outcome: Part A: Percentage of Participants With Response to Clinical Global Impression - Improvement (CGI-I) at Day 15
Description: The CGI-I employs a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. The Investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. Response choices included: 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. Higher number indicating more illness. The CGI-I is only rated at posttreatment assessments. CGI-I response were defined as having a CGI-I score "very much improved" or "much improved."
Time Frame: Day 15
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 23
percentage of participants | 47.8

12. Secondary Outcome: Part A: Insomnia Severity Index (ISI) at Day 15
Description: The ISI is a validated questionnaire designed to assess the nature, severity, and impact of insomnia. The ISI uses a 5-point Likert Scale to measure various aspects of insomnia severity (0 = none, 1 = mild, 2 = moderate; 3 = severe; 4 = very severe), satisfaction with current sleep pattern (0 = very satisfied, 1 = satisfied, 2 = neutral, 3 = dissatisfied, 4 = very dissatisfied), and various aspects of the impact of insomnia on daily functioning (0 = not at all, 1 = a little, 2 = somewhat, 3 = much, 4 = very much). ISI total score ranges from 0 to 28, where a total score of 0 to 7 = no clinically significant insomnia, 8 to 14 = subthreshold insomnia, 15 to 21 = clinical insomnia (moderate severity), and 22 to 28 = clinical insomnia (severe). A lower value indicates better outcome.
Time Frame: Day 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A (Open-label): SAGE-217
Number analyzed (Participants) | 22
score on a scale | 13.1 (6.97)

13. Secondary Outcome: Part B: Change From Baseline in the Total HAM-D Score at Day 15
Description: The 17-item HAM-D was used to rate the severity of depression in participants who were identified as experiencing an MDE. Items scored in a range of 0 to 2 include: insomnia (early, middle, late), somatic symptoms (gastrointestinal and general), genital symptoms, loss of weight, and insight. Items scored in a range of 0 to 4 include: agitation, depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), anxiety (psychic and somatic), hypochondriasis. The HAM-D total score was calculated as the sum of the 17 individual item scores, with a total score of 0 (not at all depressed) to 52 (severely depressed). Higher scores indicated more depression. A negative change from baseline indicates improvement.
Time Frame: Baseline, Day 15
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Part B: Percentage of Participants With HAM-D Response at Day 15
Description: as for outcome 7
Time Frame: Day 15
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Part B: Percentage of Participants With HAM-D Remission at Day 15
Description: as for outcome 8
Time Frame: Day 15
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Part B: Change From Baseline in the MADRS Total Score at Day 15
Description: as for outcome 9
Time Frame: Baseline, Day 15
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Part B: Change From Baseline in Response to the Clinical Global Impression - Severity (CGI-S) at Day 15
Description: as for outcome 10
Time Frame: Baseline, Day 15
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Part B: Number of Participants With Response to Clinical Global Impression - Improvement (CGI-I) at Day 15
Description: as for outcome 11
Time Frame: Day 15
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Part B: Number of Participants With At Least One Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as an adverse event with onset after the start of study through Day 42/early termination.
Time Frame: From first dose of study drug up to Day 42
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Part B: Number of Participants With TEAEs, Graded by Severity
Description: as for outcome 2
Time Frame: From first dose of study drug up to Day 42
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Part B: Percentages of Participants With Change From Baseline in Suicidal Ideation and Suicidal Behavior Based on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Suicidality was monitored using the C-SSRS. This scale consists of a baseline evaluation that assesses the lifetime experience of the participant with suicidal ideation and behavior, and a post-baseline evaluation that focuses on suicidality since the last study visit. The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) and behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt (non-fatal), completed suicide). Percentage of participants with response 'yes' were to be reported for both suicidal ideation and behavior.
Time Frame: Baseline up to Day 42
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Part B: Change From Baseline in the Young Mania Rating Scale (YMRS) Total Score
Description: as for outcome 4
Time Frame: Baseline up to Day 42
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Part B: Insomnia Severity Index (ISI) at Day 15
Description: as for outcome 12
Time Frame: Day 15
Population: Part B of the study was not conducted, so data was not collected and analyzed for this outcome measure.
Arm/Group | Part B (Double-blind): SAGE-217 | Part B (Double-blind): Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Day 42
Description: Safety Set included all participants who received at least one dose of study drug.
Arm/Group | Part A (Open-label): SAGE-217
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 10/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A (Open-label): SAGE-217 (N=35)
Somnolence (Nervous system disorders) | 4
Headache (Nervous system disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 2
Hypomania (Psychiatric disorders) | 2
Sedation (Nervous system disorders) | 2

LIMITATIONS AND CAVEATS:
Post review of Part A data, the study was stopped and, therefore, Part B was not conducted. Data was not collected or analyzed for any outcome measure planned for Part B.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-01-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT03692910/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT03692910/SAP_001.pdf